CLINICAL TRIAL: NCT06943781
Title: Research on the Application of Fecal Helicobacter Pylori Gastric Cancer Susceptibility Gene Detection in Early Diagnosis and Screening of Gastric Cancer
Brief Title: Fecal Helicobacter Pylori Gene Detection for Gastric Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Director of the gastric surgery department, Fudan University
Other Study IDs: 2410-Exp081
Record Dates: First submitted 2025-03-17; First posted 2025-04-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2024-11

CONDITIONS: Gastric Adenocarcinoma; Helicobacter Pylori

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Fecal Helicobacter pylori gastric cancer susceptibility gene test — In the early stage of the study, the team used genome-wide association analysis (GWAS) to identify H. pylori specific SNP that are significantly associated with gastric cancer in gastric cancer patients and controls; according to the mutation or not of the SNP loci, the strains were categorized into the high-risk group of gastric cancer (mutated group) and the low-risk group (un-mutated group). The mutation status of the SNP locus was detected in portable and non-invasive fecal samples from patients using molecular biology assays for early non-invasive screening and risk assessment of gastric cancer in H. pylori infected patients.

SUMMARY:
This is a prospective, multicenter, cross-sectional study. The efficacy of fecal H. pylori gastric cancer susceptibility testing in predicting gastric cancer was evaluated by comparing fecal H. pylori gastric cancer susceptibility testing with the "gold standard" imaging tests, such as CT, gastroscopy, and/or pathology, in the enrolled population.

DETAILED DESCRIPTION:
Primary study objective: to assess the sensitivity and specificity of fecal H. pylori gastric cancer susceptibility locus-based testing applied to predict gastric cancer.

Secondary research objectives: 1. the accuracy, kappa value, area under the ROC curve, positive likelihood ratio, negative likelihood ratio, positive predictive value, negative predictive value of fecal H. pylori gastric cancer susceptibility locus test applied to predict gastric cancer; 2. whether the predictive ability is significantly higher than that of the conventional tumor markers, such as CA19-9, CEA, and CA72-4, etc.; and 3. combined with fecal methylation detection Predictive ability assessment.

The "fecal H. pylori-based gastric cancer susceptibility locus test" was compared with the "gold standard" CT, gastroscopy and/or pathology, and the results were analyzed for consistency.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥40 years of age, male or female.
2. Have or will have gastroscopy and/or pathology results.
3. Have no contraindications to endoscopy and be able to cooperate with endoscopy.
4. Patients must be able to fully understand the informed consent form and be able to sign the informed consent form in person.

Exclusion Criteria:

1. Severe cardiac, hepatic, or renal insufficiency, or psychiatric disorders.
2. A previous history of upper gastrointestinal malignancy.
3. Women during pregnancy.
4. Those whose pathology is not clear.
5. Those with unsatisfactory sample retention (e.g., too small a sample size).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects for this clinical study were obtained from inpatients and outpatient follow-up patients attending the sub-centers. Subjects will be identified by the investigator based on the subject enrollment criteria and informed of the contents of the informed consent form.
  Subjects participating in the Early Diagnosis and Early Screening of Gastric Cancer study will have feces collected at the time of clinic visit or at the time of physical examination and will undergo fecal H. pylori gastric cancer susceptibility gene testing.
Sampling Method: Probability Sample
Enrollment: 13700 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
completed all phases of the study | Baseline
  The endpoint of the study will be reached if the participant has completed all phases of the study according to the study protocol (i.e., has completed sample collection, testing, and obtained "gold standard" gastroscopy and/or pathology results) or has withdrawn informed consent.

IPD SHARING:
Plan to Share IPD: Undecided